CLINICAL TRIAL: NCT05541510
Title: A Phase 2/3, Double-blind, Randomized, Placebo-controlled, 3-arm Study to Evaluate the Safety, and Efficacy of AD17002 (LTh[αK]) Intranasal Spray in Male and Female Participants Aged 18 to 65 Years With Mild to Moderate COVID 19
Brief Title: Evaluating the Safety and Efficacy of AD17002 Intranasal Spray in Treating Participants With Mild to Moderate COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The end of COVID-19 pandemic
Sponsor: Advagene Biopharma Co. Ltd. (Industry)
Collaborators: Gadjah Mada University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD17002-ID-CO
Record Dates: First submitted 2022-08-05; First posted 2022-09-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: immunomodulator; intranasal; epithelial; nasal mucosal
MeSH Terms: conditions — COVID-19 | interventions — heat-labile enterotoxin, E coli

STUDY DESIGN:
Intervention Model Description: Eligible participants confirmed for SARS-CoV-2 infection by PCR with CT values ≤28 will be randomized (1:1:1) to receive either AD17002 0 (placebo), 20, or 40 μg via the intranasal route on Days 1, 3, and 5.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Comparator (Placebo Comparator): Participants will receive placebo (formulation buffer) on treatment days 1, 3 and 5.
  Interventions: Biological: Placebo
- Low dose treatment group (Experimental): Participants will receive 20 μg of AD17002 in formulation buffer on treatment days 1, 3 and 5.
  Interventions: Biological: AD17002 + Formulation buffer
- High dose treatment group (Experimental): Participants will receive 40 μg of AD17002 in formulation buffer on treatment days 1, 3 and 5.
  Interventions: Biological: AD17002 + Formulation buffer

INTERVENTIONS:
Biological: AD17002 + Formulation buffer — Intranasal innate immune modulator
  Other Names: LTh(αK)
  Arms: High dose treatment group; Low dose treatment group
Biological: Placebo — Formulation buffer
  Other Names: Formulation buffer control
  Arms: Placebo Comparator

SUMMARY:
AD17002 enhances nasal mucosal innate immunity and has met safety and efficacy endpoints in studies of nasal adjuvants or intranasal immunomodulators. This study aims to evaluate the safety and effectiveness of AD17002 in treating patients with mild to moderate COVID-19.

All participants will be randomly divided into 1:1:1 groups and will receive standard treatment. Additionally, participants will be given either a placebo, 20, or 40 μg of AD17002 via intranasal delivery, and clinical progress will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 and ≤65 years old.
2. Laboratory confirmed SARS-CoV-2 infection, with first positive PCR test results within the past 48 hours of randomization.
3. Participants with COVID-19 symptoms within 5 days prior to the day of randomization, based on the following criteria: At least TWO of the following symptoms: Stuffy/runny nose, sore throat, shortness of breath, cough, low energy/tiredness, muscle/body aches, headache, chill/shivering, Fever (≥ 38ºC), nausea, vomiting, diarrhea, and loss of taste or smell.
4. Have a mild or moderate form of COVID-19 defined as:

   respiratory rate ≤30 breaths per minute, heart rate ≤125 beats per minute; with saturation of oxygen (SpO2) ≥93% on room air at sea level No clinical signs listed in Inclusion Criteria #3 indicative of Severe Severity
5. Have a negative pregnancy test at Screening (for female participants of childbearing potential).
6. Participant or the participant's legal representative understands the study procedures, alternative treatments available, risks involved with the study, and voluntarily agrees to participate by giving written informed consent.
7. Provide written informed consent for the study and willing to adhere to dose regimen and visit schedules.

Exclusion Criteria:

1. Participant has clinical signs suggestive of severe illnesses with SPO2≤94.
2. Sign of severe pneumonia as determined by treating physician on X-ray or SPO2
3. Participant has CT≥25 at screening
4. Participation in any other clinical study of an investigational agent treatment for SARS-CoV-2 infection within 30 days prior to the first IMP dosing.
5. Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 prior to PCR screening.
6. Participant with breakthrough SARS-CoV-2 infection within 2 weeks of SARS-CoV-2 vaccination.
7. History of severe renal disease (treatment with dialysis or phosphate binders) or clinically apparent hepatic impairment (e.g., jaundice, cholestasis, hepatic synthetic impairment, active hepatitis).
8. Impaired cardiac function or clinically significant cardiac diseases as judged by the Investigator.
9. History of anaphylaxis reaction to any known or unknown cause.
10. Immunosuppressed persons as result of illness (e.g., HIV infection) or treatment.
11. Documented history of Bell's palsy.
12. History of allergic reaction to kanamycin.
13. Immunosuppressive treatment within 3 months prior to the Screening Visit.
14. Intranasal medication or nasal topical treatment at the time of screen and study.
15. Assessed by the Investigator to be ineligible to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Time to disease improvement | [Day 1 to Day 29]
  Defined as time to achieving ≥1 decrease on WHO 11-point Clinical Progression Scale
Time to achieving the Patient Acceptable Symptom State (PASS) | [Day 1 to Day 29]
  Defined as the value of symptoms the patient considered to be well-being thresholds of the symptoms and function. The study incorporates the most widely used anchoring question to identify PASS cut-off points, which is:
  "Taking into account all your daily activities, do you consider your current state satisfactory in relation to pain level and functional impairment?" The response options were "Yes" or "No.

SECONDARY OUTCOMES:
Vital signs evaluation | [Day 1 to Day 29]
  Measuring the changes to cardiac functions
Physical examination | [Day 1 to Day 29]
  Measuring changes to physical appearances.
Clinical laboratory assessment | [Day 1 to Day 29]
  Assessing the changes to hematological parameters
Adverse events assessment | [Day 1 to Day 29]
  Adverse events graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Grade 1 (Mild) : asymptomatic or mild symptoms Grade 2 (Moderate): Local, Minimal, Moderate or noninvasive Grade 3 (Severe): Severe or medically significant but not immediately life-threatening Grade 4 (Life-threatening): Life-threatening consequences; urgent intervention indicated Grade 5 (Fatal): Death related to AE
Treatment-emergent adverse events assessment (TEAE) | [Day 1 to Day 29]
  Measuring the proportion of participants with TEAE leading to investigational medicinal products (IMPs) discontinuation.
  AE will be presented by the following categories:
  Any TEAE Treatment-related TEAE Grade 3-4, drug-related TEAE Drug-related TEAE leading to death
Nasal tolerability examination | [Day 1 to Day 29]
  Assessing the nasal symptoms by PI or delegated personnel or qualified ear, nose, and throat (ENT) specialist Symptoms include color of mucosa, turbinate swelling (middle concha and inferior concha), secretion, infection, post-nasal drip, crusting, sign of bleeding, and polyps.
Viral clearance | [Day 1 to Day 29]
  Time to clearance of SARS-CoV-2, defined as 2 consecutive negative oropharyngeal swabs by RT-PCR test and report as cycle threshold (CT)
Viral clearance rate by PCR | [Day 1 to Day 29]
  Changes of CT of RdRp (a.k.a. nsp12) N and E gene assayed by RT-PCR test
PASS evaluation | [Day 1 to Day 29]
  Proportion of subjects achieving PASS at each visit
Clinical Progression Scale analysis | [Day 1 to Day 29]
  Proportion of subjects achieving ≧1 decrease on WHO 11-point Clinical Progression Scale at each visit
Days of COVID-19 symptomatic hospitalization | [Day 1 to Day 29]
  Days participants in hospital due to infection.
Proportion of COVID-19 symptomatic hospitalization | [Day 1 to Day 29]
  Proportion of participants has been hospitalized due to infection.
Oxygen supplement treatment | [Day 1 to Day 29]
  Days of participants receive oxygen supplement.
Oxygen supplement treatment rate | [Day 1 to Day 29]
  Oxygen supplement receiving rates among infected participants
Symptom relieve days | [Day 1 to Day 29]
  Time to alleviation of each predefined COVID-19-related symptoms
Symptom severity report | [Day 1 to Day 29]
  Severity of each targeted COVID-19 symptoms An assessment of common COVID-19-related symptoms according to the FDA Guidance for Industry: Assessing COVID-19-Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment Symptom Score Guide: 0= None; 1= Mild; 2= Moderately; 3= Severe
Mortality rate report | [Day 1 to Day 29]
  Proportion of participants with death (all cause)

OTHER OUTCOMES:
Anti-SARS-CoV-2 specific IgG assessment | [Day 1 and Day 29]
  The titers of anti-SARS-CoV-2 specific IgG of each participants are measured with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Jarir At Thobari, MD. PhD., Study Chair — Gadjah Mada University
Locations (3):
- Indonesia (3):
  - RSPI Sulianti Saroso, Kota Jkt Utara, DKI Jakarta
  - RSDC Wisma Atlit, Kota Jkt Utara, DKI Jakarta
  - RSA UGM, Yogyakarta, Special Region of Yogyakarta